CLINICAL TRIAL: NCT01557322
Title: Evaluation of the Clinical Characteristics, Real-world Treatment Pathways, and Outcomes of Patients With Moderate Rheumatoid Arthritis
Brief Title: Characterize Patients With Moderately Active Rheumatoid Arthritis (RA)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1801345
Record Dates: First submitted 2012-02-08; First posted 2012-03-19 (Estimated); Results first posted 2013-10-31 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept; Methotrexate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Biologic
  Interventions: Biological: etanercept
- non-biologic DMARD
  Interventions: Drug: methotrexate (MTX)

INTERVENTIONS:
Biological: etanercept — This is a Non-interventional study. The data is being analyzed retrospectively. The data consists of 2 cohorts; biologic and non-biologic
  Other Names: Enrel
  Groups: Biologic
Drug: methotrexate (MTX) — This is a Non-interventional study. The data is being analyzed retrospectively. The data consists of 2 cohorts; biologic and non-biologic
  Other Names: non-biologic DMARD
  Groups: non-biologic DMARD

SUMMARY:
1. To assess the baseline (i.e. RA therapy initiation) characteristics in a real-world setting across two moderate RA cohorts: a Test Group of patients newly exposed to etanercept (Enbrel) therapy and a Control Group of patients with similar disease characteristics newly exposed to other, non-biologic therapies.
2. To assess the change over time (from baseline to the most recent follow-up) in the characteristics described at baseline in 2 British Society for Rheumatology Biologics Register (BSRBR) cohorts (i.e. moderate RA patients treated with Disease modifying anti-rheumatic drugs (DMARDs) alone versus moderate RA patients treated with Enbrel).

DETAILED DESCRIPTION:
Retrospective database analysis

ELIGIBILITY:
Inclusion Criteria:

The Test Group will be patients with rheumatoid arthritis, newly starting therapy with etanercept (Enbrel). Inclusion criteria for the exposed cohort subjects are:

* Patients aged 18 years and over at the time of diagnosis;
* Patients from the BSRBR with moderate RA as defined by a DAS28 (>3.2 and ≤5.1);
* Patients who have given informed consent for long term follow-up and access to all medical records;
* Patients initiating (i.e. at leats one treatment) treatment with etanercept (Enbrel) for RA.

The Control Group:

* Patients aged 18 years and over a the time of diagnosis;
* Patients from the BSRBR with moderate RA as defined by a DAS28 (>3.2 and ≤5.1);
* Patients who have given informed consent for long term follow-up and access to all medical records; Patients are receiving at least one traditional DMARD and have never been prescribed a biologic agent;

Exclusion Criteria:

Per BSRBR registry since data is retropsectively being analyzed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The BSR Biologics Register tracks the progress of patients with severe rheumatoid arthritis and other rheumatic conditions who are taking biologic therapy and those who are biologic naive.
Sampling Method: Non-Probability Sample
Enrollment: 1754 (Actual)
Dates: Start 2011-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1801345&StudyName=Characterize%20Patients%20with%20Moderately%20Active%20Rheumatoid%20Arthritis%20%28RA%29

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept: Participants with moderate rheumatoid arthritis (RA), defined as disease activity score based on 28-joints count (DAS28) more than (>) 3.2 to less than or equal to (<=) 5.1, who received etanercept (ETN, as their first biological drug) in doses as per approved product label or summary of product characteristics (SmPC), were followed retrospectively using the data in British Society for Rheumatology Biologics Register (BSRBR) for 5 years. The doses had been adjusted according to medical and therapeutic necessity.
- nbDMARDs: Biological naïve participants with moderate RA, defined as DAS28 >3.2 to <=5.1, who received non-biologic disease modifying anti-rheumatic drugs (nbDMARDs) in doses as per approved product label or SmPC, were followed retrospectively using the data in BSRBR for 5 years. The doses had been adjusted according to medical and therapeutic necessity.
Period: Overall Study
Arm/Group | Etanercept | nbDMARDs
Started | 211 | 1543
Completed | 211 | 1543
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Etanercept | nbDMARDs | Total
Number analyzed (Participants) | 211 | 1543 | 1754
Age Continuous [Median (Full Range); unit: years] | 55.3 [18.9 to 81.0] | 62.1 [18.2 to 86.7] | 61.2 [18.2 to 86.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 163 | 1098 | 1261
  Male | 48 | 445 | 493

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With American College of Rheumatology (ACR) Criteria
Description: ACR criteria: 1) Morning stiffness: in and around joints, lasting at least (>=) 1 hour; 2) Arthritis/deformity of >=3 joint areas: presence of soft tissue swelling or fluid (not bony overgrowth alone), 14 possible areas are right/left proximal interphalangeal (PIP), metacarpophalangeal (MCP), wrist, elbow, knee, ankle, metatarsophalangeal (MTP) joints; 3) Arthritis of hand joints: >=1 area swollen in wrist, MCP, PIP joint; 4) Symmetric arthritis: simultaneous involvement of same joint areas (as defined in 2) on both sides of body; 5): Rheumatoid nodules: subcutaneous nodules over bony prominences or extensor surfaces or in juxtaarticular regions; 6): Rheumatoid factor (RF): abnormal amounts of RF by any method for which result has been positive in <5% of normal control participants; 7) Radiographic changes: typical of RA on posteroanterior hand and wrist radiographs, which must include erosions/unequivocal bony decalcification localized in or most marked adjacent to involved joints.
Time Frame: Baseline
Population: Analysis population included all enrolled participants with moderate RA at baseline. Here "N" (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 211 | 1541
participants
  Morning Stiffness >1 Hour | 194 | 1316
  Arthritis/Deformity of >=3 Joint Areas | 179 | 1133
  Arthritis/Deformity of Hand/Joint | 160 | 1123
  Symmetry | 175 | 978
  Nodules | 91 | 470
  Rheumatoid Factor Positive | 123 | 927
  Erosions on Hand or Feet X-Ray | 116 | 730
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; Morning Stiffness > 1 Hour: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.010, Chi-squared
Statistical Analysis 2: Comparison: Etanercept vs nbDMARDs; Arthritis or Deformity of 3 or More Joint Areas: p-value was calculated using chi-square test; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 3: Comparison: Etanercept vs nbDMARDs; Arthritis/Deformity of Hand/Joint: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.363, Chi-squared
Statistical Analysis 4: Comparison: Etanercept vs nbDMARDs; Symmetry: p-value was calculated using chi-square test; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 5: Comparison: Etanercept vs nbDMARDs; Nodules: p-value was calculated using chi-square test; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 6: Comparison: Etanercept vs nbDMARDs; Rheumatoid Factor Positive: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.605, Chi-squared
Statistical Analysis 7: Comparison: Etanercept vs nbDMARDs; Erosions on Hand or Feet X-Ray: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.038, Chi-squared

2. Primary Outcome: Number of Participants With Systemic Features
Description: Systemic features included sicca syndrome, serosal involvement (pleurisy/pericarditis), eye involvement, systemic vasculitis, nailfold vasculitis, pulmonary fibrosis, and others (other than those specified).
Time Frame: Baseline
Population: Analysis population included all enrolled participants with moderate RA at baseline. Here "N" (number of participants analyzed) signifies participants who were evaluable for this measure and "n" signifies participants evaluable for specified category for each treatment arm, respectively.
Measure: Number; unit: participants
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 211 | 1540
participants
  Sicca Syndrome (n= 211, 1540) | 45 | 166
  Serosal Involvement (n= 211, 1540) | 7 | 18
  Eye Involvement (n= 211, 1540) | 17 | 93
  Systemic Vasculitis (n= 211, 1540) | 6 | 14
  Nailfold Vasculitis (n= 211, 1540) | 3 | 17
  Pulmonary Fibrosis (n= 211, 1540) | 2 | 37
  Other (n= 211, 1537) | 6 | 34
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; Sicca Syndrome: p-value was calculated using chi-square test; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: Etanercept vs nbDMARDs; Serosal Involvement: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.024, Chi-squared
Statistical Analysis 3: Comparison: Etanercept vs nbDMARDs; Eye Involvement: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.257, Chi-squared
Statistical Analysis 4: Comparison: Etanercept vs nbDMARDs; Systemic Vasculitis: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.026, Chi-squared
Statistical Analysis 5: Comparison: Etanercept vs nbDMARDs; Nailfold Vasculitis: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.725, Chi-squared
Statistical Analysis 6: Comparison: Etanercept vs nbDMARDs; Pulmonary Fibrosis: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.220, Chi-squared
Statistical Analysis 7: Comparison: Etanercept vs nbDMARDs; Other: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.620, Chi-squared

3. Primary Outcome: Number of Participants With Prior Joint Replacement or Surgery
Description: Participants who had prior total knee replacement, total hip replacement, total shoulder replacement, total elbow replacement, wrist/hand/ankle/foot surgery, and neck surgery are reported.
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 211 | 1540
participants
  Total Knee Replacement | 31 | 141
  Total Hip Replacement | 29 | 99
  Total Shoulder Replacement | 21 | 24
  Total Elbow Replacement | 14 | 31
  Wrist/Hand/Ankle/Foot Surgery | 56 | 262
  Neck Surgery | 9 | 9
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; Total Knee Replacement: p-value was calculated using chi-square test; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: Etanercept vs nbDMARDs; Total Hip Replacement: p-value was calculated using chi-square test; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 3: Comparison: Etanercept vs nbDMARDs; Total Shoulder Replacement: p-value was calculated using chi-square test; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 4: Comparison: Etanercept vs nbDMARDs; Total Elbow Replacement: p-value was calculated using chi-square test; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 5: Comparison: Etanercept vs nbDMARDs; Wrist/Hand/Ankle/Foot Surgery: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.001, Chi-squared
Statistical Analysis 6: Comparison: Etanercept vs nbDMARDs; Neck Surgery: p-value was calculated using chi-square test; Test type: Superiority or Other; p < 0.001, Chi-squared

4. Primary Outcome: Number of Participants With Chest X-Ray Prior to New Therapy
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 194 | 1441
participants | 183 | 742
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; P-value was calculated using chi-square test; Test type: Superiority or Other; p < 0.001, Chi-squared

5. Primary Outcome: Number of Participants With Comorbidities
Description: Comorbidities included: hypertension, moderate or severe heart failure, angina, stroke, epilepsy, asthma, chronic bronchitis/emphysema, peptic ulcer, tuberculosis, pre-existing or recent onset of central nervous system demyelinating disorders, chronic infectious disease such as chronic renal infection, chronic chest infection with bronchiectasis or sinusitis, active tuberculosis, renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic or cerebral disease, malignancy or history of malignancy, hyperthyroidism, depression and/or anxiety, recent substance abuse (drug or alcohol), human immunodeficiency virus (HIV) infection or active hepatitis B/C infection (including associated chronic active hepatitis). Participants suffering from any of the comorbidity are reported.
Time Frame: Baseline
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 208 | 1541
participants
  High Blood Pressure (n= 208, 1532) | 60 | 488
  Angina (n= 211, 1536) | 5 | 115
  Heart Attack (n= 210, 1535) | 6 | 73
  Stroke (n= 211, 1538) | 3 | 53
  Epilepsy (n= 211, 1541) | 2 | 19
  Asthma (n= 211, 1539) | 24 | 198
  Chronic Bronchitis/Emphysema (n= 211, 1537) | 8 | 124
  Peptic Ulcer (n= 208, 1537) | 11 | 97
  Liver Disease (n= 211, 1539) | 11 | 26
  Renal Disease (n= 211, 1540) | 8 | 46
  Tuberculosis (n= 207, 1538) | 5 | 34
  Demyelination (n= 210, 1536) | 1 | 7
  Diabetes (n= 211, 1539) | 16 | 93
  Hyperthyroidism (n= 211, 1535) | 3 | 65
  Depression (n= 211, 1539) | 40 | 249
  Cancer (n= 210, 1540) | 6 | 102
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; High Blood Pressure: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.381, Chi-squared
Statistical Analysis 2: Comparison: Etanercept vs nbDMARDs; Angina: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.006, Chi-squared
Statistical Analysis 3: Comparison: Etanercept vs nbDMARDs; Heart Attack: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.215, Chi-squared
Statistical Analysis 4: Comparison: Etanercept vs nbDMARDs; Stroke: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.117, Chi-squared
Statistical Analysis 5: Comparison: Etanercept vs nbDMARDs; Epilepsy: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 1.000, Chi-squared
Statistical Analysis 6: Comparison: Etanercept vs nbDMARDs; Asthma: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.542, Chi-squared
Statistical Analysis 7: Comparison: Etanercept vs nbDMARDs; Chronic Bronchitis/Emphysema: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.027, Chi-squared
Statistical Analysis 8: Comparison: Etanercept vs nbDMARDs; Peptic Ulcer: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.566, Chi-squared
Statistical Analysis 9: Comparison: Etanercept vs nbDMARDs; Liver Disease: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.003, Chi-squared
Statistical Analysis 10: Comparison: Etanercept vs nbDMARDs; Renal Disease: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.526, Chi-squared
Statistical Analysis 11: Comparison: Etanercept vs nbDMARDs; Tuberculosis: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.802, Chi-squared
Statistical Analysis 12: Comparison: Etanercept vs nbDMARDs; Demyelination: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 1.000, Chi-squared
Statistical Analysis 13: Comparison: Etanercept vs nbDMARDs; Diabetes: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.385, Chi-squared
Statistical Analysis 14: Comparison: Etanercept vs nbDMARDs; Hyperthyroidism: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.048, Chi-squared
Statistical Analysis 15: Comparison: Etanercept vs nbDMARDs; Depression: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.308, Chi-squared
Statistical Analysis 16: Comparison: Etanercept vs nbDMARDs; Cancer: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.033, Chi-squared

6. Primary Outcome: Body Mass Index (BMI)
Description: BMI was calculated by weight divided by height squared and measured as kilogram per square meter (kg/m^2).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 178 | 1462
kg/m^2 | 26.6 (0.4) | 27.2 (0.1)
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; P-value was calculated using 2-sided t-test; Test type: Superiority or Other; p = 0.188, t-test, 2 sided

7. Primary Outcome: Blood Pressure (BP)
Description: BP is the pressure of the blood within the arteries. It is produced primarily by the contraction of the heart muscle. BP measurement is recorded by 2 numbers: systolic BP (SBP, BP when heart is contracting; it is the maximum arterial pressure during contraction of left ventricle) and diastolic BP (DBP, BP when heart is relaxing; it is the minimum arterial pressure during relaxation and dilation of ventricles).
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Error); unit: millimeter of mercury (mmHg)
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 199 | 1483
millimeter of mercury (mmHg)
  Systolic Blood Pressure (n= 199, 1477) | 134.3 (1.4) | 138.0 (0.5)
  Diastolic Blood Pressure (n= 199, 1483) | 79.4 (0.8) | 80.2 (0.3)
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; Systolic Blood Pressure: p-value was calculated using 2-sided t-test; Test type: Superiority or Other; p = 0.016, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs nbDMARDs; Diastolic Blood Pressure: p-value was calculated using 2-sided t-test; Test type: Superiority or Other; p = 0.369, t-test, 2 sided

8. Primary Outcome: Change From Baseline in Disease Activity Score Based on 28-joints Count (DAS28) at Month 60
Description: DAS28 calculated from the number of swollen joints (SJC) and painful joints (PJC) using the 28 joints count, acute phase reactants (erythrocyte sedimentation rate [ESR, millimeters per hour] or C-reactive protein [CRP, milligram per liter]) and patient's global assessment (PtGA) of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). DAS28 <2.6: remission, DAS28 <=3.2: low disease activity, DAS28 >3.2 to <=5.1: moderate disease activity, DAS28 >5.1: progression.
Time Frame: Baseline, Month 60
Population: Analysis population included all enrolled participants with moderate RA at baseline. Here "n" signifies participants evaluable at each time-point for each treatment arm, respectively.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 211 | 1543
units on a scale
  Baseline (n= 211, 1543) | 4.6 (0.03) | 4.4 (0.01)
  Change at Month 60 (n= 57, 131) | -1.67 (0.55) | -1.45 (0.55)
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; Baseline: p-value was calculated using 2-sided t-test; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs nbDMARDs; Change at Month 60: p-value was calculated using multivariate linear regression with baseline DAS28 score and other baseline variables (socio-demographics, disease characteristics, and initial treatment profile) as covariates; Test type: Superiority or Other; p = 0.3746, Regression, Linear

9. Primary Outcome: Change From Baseline in Tender Joints Count (TJC) at Month 60
Description: Number of tender joints was determined by examining 28 joints and identified the joints that were painful under pressure or to passive motion. The number of tender joints was recorded on the joint assessment form at each visit, no tenderness = 0, tenderness = 1. A negative value in change from baseline indicates an improvement.
Time Frame: Baseline, Month 60
Population: Analysis population included all enrolled participants with moderate RA at baseline. Here "N" (number of participants analyzed) signifies participants who were evaluable for this measure and "n" signifies participants evaluable at each time-point for each treatment arm, respectively.
Measure: Mean (Standard Error); unit: tender joints
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 207 | 1526
tender joints
  Baseline (n= 207, 1526) | 6.1 (0.3) | 4.8 (0.1)
  Change at Month 60 (n= 55, 2) | NA (NA) — Result not reported as there was insufficient data to evaluate the effect in multivariate model. | NA (NA) — Result not reported as there was insufficient data to evaluate the effect in multivariate model.
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; Baseline: p-value was calculated using 2-sided t-test; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

10. Primary Outcome: Change From Baseline in Swollen Joints Count (SJC) at Month 60
Description: Number of swollen joints was determined by examination of 28 joints and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form at each visit, no swelling = 0, swelling =1. A negative value in change from baseline indicates an improvement.
Time Frame: Baseline, Month 60
Population: as for outcome 9
Measure: Mean (Standard Error); unit: swollen joints
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 206 | 1526
swollen joints
  Baseline (n= 206, 1526) | 6.0 (0.4) | 3.8 (0.1)
  Change at Month 60 (n= 55, 2) | NA (NA) — Result not reported as there was insufficient data to evaluate the effect in multivariate model. | NA (NA) — Result not reported as there was insufficient data to evaluate the effect in multivariate model.
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; Baseline: p-value was calculated using 2-sided t-test; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

11. Primary Outcome: Change From Baseline in C-Reactive Protein (CRP) Level at Month 60
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultra-sensitive assay. Normal range of CRP is <10 milligram/liter (mg/L). A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline, Month 60
Population: as for outcome 9
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 80 | 431
mg/L
  Baseline (n= 80, 431) | 28.3 (3.4) | 23.1 (1.4)
  Change at Month 60 (n= 15, 0) | NA (NA) — Result not reported as there was insufficient data to evaluate the effect in multivariate model. | NA (NA) — Result not reported as no participants were evaluable at this time-point.
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; Baseline: p-value was calculated using 2-sided t-test; Test type: Superiority or Other; p = 0.154, t-test, 2 sided

12. Primary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate (ESR) at Month 60
Description: ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube. Normal range is 0-30 millimeter/hour (mm/hr). A higher rate is consistent with inflammation.
Time Frame: Baseline, Month 60
Population: as for outcome 9
Measure: Mean (Standard Error); unit: mm/hour
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 200 | 134
mm/hour
  Baseline (n= 200, 1344) | 24.0 (1.3) | 26.3 (0.5)
  Change at Month 60 (n= 53, 7) | NA (NA) — Result not reported as there was insufficient data to evaluate the effect in multivariate model. | NA (NA) — Result not reported as there was insufficient data to evaluate the effect in multivariate model.
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; Baseline: p-value was calculated using 2-sided t-test; Test type: Superiority or Other; p = 0.108, t-test, 2 sided

13. Primary Outcome: Change From Baseline in Patient's Global Assessment (PtGA) of Disease Activity at Month 60
Description: Participants answered: "Considering all the ways your arthritis affects you, how are you feeling today?" Participants responded by using a 0 - 100 mm VAS, where 0 mm = very well and 100 mm = very poorly.
Time Frame: Baseline, Month 60
Population: as for outcome 9
Measure: Mean (Standard Error); unit: mm
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 205 | 1525
mm
  Baseline (n= 205, 1525) | 49.0 (1.7) | 46.7 (0.5)
  Change at Month 60 (n= 53, 2) | NA (NA) — Result not reported as there was insufficient data to evaluate the effect in multivariate model. | NA (NA) — Result not reported as there was insufficient data to evaluate the effect in multivariate model.
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; Baseline: p-value was calculated using 2-sided t-test; Test type: Superiority or Other; p = 0.199, t-test, 2 sided

14. Primary Outcome: Duration of Disease (Rheumatoid Arthritis)
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Error); unit: years
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 208 | 1529
years | 14.1 (0.7) | 10.2 (0.3)
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; P-value was calculated using 2-sided t-test; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

15. Primary Outcome: Time Since First Rheumatologist Visit
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Error); unit: years
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 204 | 1501
years | 13.1 (0.7) | 9.7 (0.3)
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; P-value was calculated using 2-sided t-test; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

16. Primary Outcome: Time Since Recalled Symptom Onset
Description: RA symptoms include joint pain, stiffness, and swelling.
Time Frame: Baseline
Population: Results not reported as this outcome was not evaluated due to lack availability of information on the outcome in BSRBR used for analysis.
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 0 | 0

17. Primary Outcome: Number of Participants With Previous and Current Disease Modifying Anti-Rheumatic Drugs (DMARDs)
Description: Number of participants who previously received DMARDs or were currently on DMARDs at baseline is reported.
Time Frame: Baseline
Population: Analysis population included all enrolled participants with moderate RA at baseline.
Measure: Number; unit: participants
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 211 | 1543
participants
  Current DMARDs: Methotrexate | 65 | 963
  Current DMARDs: Azathioprine | 7 | 32
  Current DMARDs: Cyclophosphamide | 0 | 2
  Current DMARDs: Cyclosporine | 0 | 27
  Current DMARDs: Leflunomide | 14 | 158
  Current DMARDs: Sulphasalazine | 20 | 370
  Previous DMARDs: Methotrexate | 198 | 1158
  Previous DMARDs: Azathioprine | 61 | 118
  Previous DMARDs: Cyclophosphamide | 10 | 7
  Previous DMARDs: Cyclosporine | 40 | 70
  Previous DMARDs: Leflunomide | 111 | 209
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; Current DMARDs, Methotrexate: p-value was calculated using chi-square test; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: Etanercept vs nbDMARDs; Current DMARDs, Azathioprine: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.313, Chi-squared
Statistical Analysis 3: Comparison: Etanercept vs nbDMARDs; Current DMARDs, Cyclophosphamide: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 1.000, Chi-squared
Statistical Analysis 4: Comparison: Etanercept vs nbDMARDs; Current DMARDs, Cyclosporine: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.066, Chi-squared
Statistical Analysis 5: Comparison: Etanercept vs nbDMARDs; Current DMARDs, Leflunomide: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.099, Chi-squared
Statistical Analysis 6: Comparison: Etanercept vs nbDMARDs; Current DMARDs, Sulphasalazine: p-value was calculated using chi-square test; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 7: Comparison: Etanercept vs nbDMARDs; Previous DMARDs, Methotrexate: p-value was calculated using chi-square test; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 8: Comparison: Etanercept vs nbDMARDs; Previous DMARDs, Azathioprine: p-value was calculated using chi-square test; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 9: Comparison: Etanercept vs nbDMARDs; Previous DMARDs, Cyclophosphamide: p-value was calculated using chi-square test; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 10: Comparison: Etanercept vs nbDMARDs; Previous DMARDs, Cyclosporine: p-value was calculated using chi-square test; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 11: Comparison: Etanercept vs nbDMARDs; Previous DMARDs, Leflunomide: p-value was calculated using chi-square test; Test type: Superiority or Other; p < 0.001, Chi-squared

18. Primary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) Score at Month 60
Description: Health Assessment Questionnaire-Disability Index (HAQ-DI): participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0 = no difficulty; 1 = some difficulty; 2 = much difficulty; 3 = unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0 to 3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Baseline, Month 60
Population: as for outcome 9
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 195 | 1294
units on a scale
  Baseline (n= 195, 1294) | 1.9 (0.07) | 1.5 (0.04)
  Change at Month 60 (n= 0, 0) | NA (NA) — Result not reported as no participants were evaluable at this time-point. | NA (NA) — Result not reported as no participants were evaluable at this time-point.
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; Baseline: p-value was calculated using 2-sided t-test; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

19. Primary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) at Month 60
Description: The 36-Item Short-Form Health Survey (SF-36) is a standardized survey evaluating 8 aspects of functional health and well-being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. These 8 aspects can also be summarized as physical component score (PCS) and mental component score (MCS). Total of 3 variables were analyzed (2 composite subscales and vitality score). The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning).
Time Frame: Baseline, Month 60
Population: as for outcome 9
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 186 | 1272
units on a scale
  Baseline: PCS (n= 171, 1202) | 27.3 (0.5) | 29.8 (0.2)
  Baseline: MCS (n= 171, 1202) | 49.1 (0.6) | 49.2 (0.2)
  Baseline: Vitality Score (n= 186, 1272) | 49.2 (0.5) | 49.0 (0.2)
  Change at Month 60: PCS (n= 0, 0) | NA (NA) — Result not reported as no participants were evaluable at this time-point. | NA (NA) — Result not reported as no participants were evaluable at this time-point.
  Change at Month 60: MCS (n= 0, 0) | NA (NA) — Result not reported as no participants were evaluable at this time-point. | NA (NA) — Result not reported as no participants were evaluable at this time-point.
  Change at Month 60: Vitality Score (n= 0, 0) | NA (NA) — Result not reported as no participants were evaluable at this time-point. | NA (NA) — Result not reported as no participants were evaluable at this time-point.
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; Baseline PCS: p-value was calculated using 2-sided t-test; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs nbDMARDs; Baseline MCS: p-value was calculated using 2-sided t-test; Test type: Superiority or Other; p = 0.886, t-test, 2 sided
Statistical Analysis 3: Comparison: Etanercept vs nbDMARDs; Baseline Vitality Score: p-value was calculated using 2-sided t-test; Test type: Superiority or Other; p = 0.680, t-test, 2 sided

20. Primary Outcome: Change From Baseline in Euro Quality of Life - 5 Dimensions (EQ-5D) at Month 60
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state (confined to bed). Scoring formula developed by EuroQoL Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Baseline, Month 60
Population: Data not analyzed due to low number of participants available for this measure in BSRBR used for analysis.
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 0 | 0

21. Primary Outcome: Time to Disease Worsening
Description: Disease worsening (severe RA diagnosis) was defined as DAS28 score >5.1.
Time Frame: Baseline up to Month 60
Population: Data not analyzed due to low number of participants available for this measure in BSRBR used for analysis.
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 0 | 0

22. Primary Outcome: Time to Therapeutic Goal
Description: Therapeutic goal achievement was based on physician's discretion.
Time Frame: Baseline up to Month 60
Population: Data not analyzed due to low number of participants available for this measure in BSRBR used for analysis.
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 0 | 0

23. Primary Outcome: Change From Baseline in Pain Visual Analog Scale (VAS) Score at Month 60
Description: The pain VAS is a horizontal line; 100 millimeter (mm) in length, self-administered by the participant to rate pain from 0 mm (no pain) to 100 mm (worst possible pain).Change = mean scores at observation minus mean scores at baseline.
Time Frame: Baseline, Month 60
Population: Data not analyzed due to low number of participants available for this measure in BSRBR used for analysis.
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 0 | 0

24. Primary Outcome: Number of Participants Achieving American College of Rheumatology 20% (ACR20) Response at Month 60
Description: ACR20 response: greater than or equal to (>=) 20 percent (%) improvement in tender joints count (TJC); >= 20% improvement in swollen joints count (SJC); and >= 20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP).
Time Frame: Month 60
Population: Result not reported as no participants were evaluable at this time-point.
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 0 | 0

25. Primary Outcome: Number of Participants Achieving American College of Rheumatology 50% (ACR50) Response at Month 60
Description: ACR50 response: >= 50% improvement in TJC or SJC and 50% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Month 60
Population: Result not reported as no participants were evaluable at this time-point.
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 0 | 0

26. Primary Outcome: Number of Participants Achieving American College of Rheumatology 70% (ACR70) Response at Month 60
Description: ACR70 response: >=70% improvement in TJC or SJC and 70% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Month 60
Population: Result not reported as no participants were evaluable at this time-point.
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 0 | 0

27. Primary Outcome: Number of Rheumatoid Arthritis (RA) Related Visits
Description: Number of RA-related visits to doctor/healthcare professional in previous 3 months was to be reported.
Time Frame: Baseline
Population: Results not reported as this outcome was not evaluated due to lack of availability of information on the outcome in BSRBR used for analysis.
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 0 | 0

28. Primary Outcome: Direct and Indirect Cost of Rheumatoid Arthritis (RA) Treatment
Description: Direct costs included: outpatient costs, physician visits, outpatient surgery, emergency room visits, visits to healthcare professionals other than physicians, medications, diagnostic and/or therapeutic procedures, medical devices, inpatient costs, admission to acute-care nonsurgical departments, admission to acute-care surgical departments, admission to extended-care facilities, and other direct costs (travel expenses, home care, home remodeling, medical devices, non-physician healthcare professionals, alternative medicine practitioner, participant time). Indirect cost (related to lost productivity through morbidity and death) included: lost productivity in employed participants (disability, sick-leaves), lost opportunities (lost productivity in family members caring for the patient, disability requiring changes to everyday activities), and lost wages.
Time Frame: Baseline
Population: as for outcome 27
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 0 | 0

29. Other Pre Specified Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Number of participants with AEs is reported by each follow-up time point up to Month 60.
Time Frame: Month 6, 12, 18, 24, 30, 36, 48, 60
Population: Analysis population included all enrolled participants with moderate RA at baseline.
Measure: Number; unit: participants
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 211 | 1543
participants
  Month 6 | 22 | 101
  Month 12 | 10 | 100
  Month 18 | 12 | 111
  Month 24 | 10 | 102
  Month 30 | 12 | 80
  Month 36 | 6 | 91
  Month 48 | 3 | 63
  Month 60 | 7 | 44
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; Month 6: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.0233, Chi-squared
Statistical Analysis 2: Comparison: Etanercept vs nbDMARDs; Month 12: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.5103, Chi-squared
Statistical Analysis 3: Comparison: Etanercept vs nbDMARDs; Month 18: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.9990, Chi-squared
Statistical Analysis 4: Comparison: Etanercept vs nbDMARDs; Month 24: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.6495, Chi-squared
Statistical Analysis 5: Comparison: Etanercept vs nbDMARDs; Month 30: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.3829, Chi-squared
Statistical Analysis 6: Comparison: Etanercept vs nbDMARDs; Month 36: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.1085, Chi-squared
Statistical Analysis 7: Comparison: Etanercept vs nbDMARDs; Month 48: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.0472, Chi-squared
Statistical Analysis 8: Comparison: Etanercept vs nbDMARDs; Month 60: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.4804, Chi-squared

30. Other Pre Specified Outcome: Number of Participants With Malignancy
Description: Malignancy included lymphoproliferative tumors, Hodgkins lymphoma, myeloma, leukaemia, non-melanoma skin cancer, and solid tumor. Number of participants with each of these malignancies is reported by each follow-up time point up to Month 60.
Time Frame: Month 6, 12, 18, 24, 30, 36, 48, 60
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 191 | 1457
participants
  Lymphoproliferative Tumors: Month 6 (n=191, 1457) | 1 | 1
  Lymphoproliferative Tumors: Month 12 (n=172, 1394) | 1 | 1
  Lymphoproliferative Tumors: Month 18 (n=146, 1350) | 1 | 0
  Lymphoproliferative Tumors: Month 24 (n=141, 1245) | 0 | 0
  Lymphoproliferative Tumors: Month 30 (n=127, 1097) | 0 | 3
  Lymphoproliferative Tumors: Month 36 (n=128, 1027) | 1 | 1
  Lymphoproliferative Tumors: Month 48 (n=114, 815) | 1 | 0
  Lymphoproliferative Tumors: Month 60 (n=108, 516) | 0 | 0
  Hodgkins Lymphoma: Month 6 (n=191, 1457) | 1 | 1
  Hodgkins Lymphoma: Month 12 (n=172, 1394) | 0 | 0
  Hodgkins Lymphoma: Month 18 (n=146, 1350) | 1 | 0
  Hodgkins Lymphoma: Month 24 (n=141, 1245) | 0 | 0
  Hodgkins Lymphoma: Month 30 (n=127, 1097) | 0 | 2
  Hodgkins Lymphoma: Month 36 (n=128, 1027) | 1 | 1
  Hodgkins Lymphoma: Month 48 (n=114, 815) | 1 | 0
  Hodgkins Lymphoma: Month 60 (n=108, 516) | 0 | 0
  Myeloma: Month 6 (n=191, 1457) | 0 | 0
  Myeloma: Month 12 (n=172, 1394) | 0 | 1
  Myeloma: Month 18 (n=146, 1350) | 0 | 0
  Myeloma: Month 24 (n=141, 1245) | 0 | 0
  Myeloma: Month 30 (n=127, 1097) | 0 | 1
  Myeloma: Month 36 (n=128, 1027) | 0 | 0
  Myeloma: Month 48 (n=114, 815) | 0 | 0
  Myeloma: Month 60 (n=108, 516) | 0 | 0
  Leukaemia: Month 6 (n=191, 1457) | 0 | 0
  Leukaemia: Month 12 (n=172, 1394) | 1 | 0
  Leukaemia: Month 18 (n=146, 1350) | 0 | 0
  Leukaemia: Month 24 (n=141, 1245) | 0 | 0
  Leukaemia: Month 30 (n=127, 1097) | 0 | 0
  Leukaemia: Month 36 (n=128, 1027) | 0 | 0
  Leukaemia: Month 48 (n=114, 815) | 0 | 0
  Leukaemia: Month 60 (n=108, 516) | 0 | 0
  Non-Melanoma Skin Cancer: Month 6 (n=191, 1457) | 0 | 5
  Non-Melanoma Skin Cancer: Month 12 (n=172, 1394) | 0 | 6
  Non-Melanoma Skin Cancer: Month 18 (n=146, 1350) | 0 | 4
  Non-Melanoma Skin Cancer: Month 24 (n=141, 1245) | 1 | 9
  Non-Melanoma Skin Cancer: Month 30 (n=127, 1097) | 0 | 4
  Non-Melanoma Skin Cancer: Month 36 (n=128, 1027) | 0 | 3
  Non-Melanoma Skin Cancer: Month 48 (n=114, 815) | 0 | 6
  Non-Melanoma Skin Cancer: Month 60 (n=108, 516) | 0 | 0
  Solid Tumor: Month 6 (n=191, 1457) | 2 | 9
  Solid Tumor: Month 12 (n=172, 1394) | 0 | 4
  Solid Tumor: Month 18 (n=146, 1350) | 0 | 9
  Solid Tumor: Month 24 (n=141, 1245) | 0 | 4
  Solid Tumor: Month 30 (n=127, 1097) | 2 | 5
  Solid Tumor: Month 36 (n=128, 1027) | 0 | 7
  Solid Tumor: Month 48 (n=114, 815) | 2 | 5
  Solid Tumor: Month 60 (n=108, 516) | 0 | 3
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; Lymphoproliferative Tumors, Month 6: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.0895, Chi-squared
Statistical Analysis 2: Comparison: Etanercept vs nbDMARDs; Lymphoproliferative Tumors, Month 12: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.0774, Chi-squared
Statistical Analysis 3: Comparison: Etanercept vs nbDMARDs; Lymphoproliferative Tumors, Month 18: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.0024, Chi-squared
Statistical Analysis 4: Comparison: Etanercept vs nbDMARDs; Lymphoproliferative Tumors, Month 30: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.5552, Chi-squared
Statistical Analysis 5: Comparison: Etanercept vs nbDMARDs; Lymphoproliferative Tumors, Month 36: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.0793, Chi-squared
Statistical Analysis 6: Comparison: Etanercept vs nbDMARDs; Lymphoproliferative Tumors, Month 48: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.0075, Chi-squared
Statistical Analysis 7: Comparison: Etanercept vs nbDMARDs; Hodgkins Lymphoma, Month 6: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.0895, Chi-squared
Statistical Analysis 8: Comparison: Etanercept vs nbDMARDs; Hodgkins Lymphoma, Month 18: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.0024, Chi-squared
Statistical Analysis 9: Comparison: Etanercept vs nbDMARDs; Hodgkins Lymphoma, Month 30: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.6301, Chi-squared
Statistical Analysis 10: Comparison: Etanercept vs nbDMARDs; Hodgkins Lymphoma, Month 36: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.0793, Chi-squared
Statistical Analysis 11: Comparison: Etanercept vs nbDMARDs; Hodgkins Lymphoma, Month 48: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.0075, Chi-squared
Statistical Analysis 12: Comparison: Etanercept vs nbDMARDs; Myeloma, Month 12: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.7253, Chi-squared
Statistical Analysis 13: Comparison: Etanercept vs nbDMARDs; Myeloma, Month 30: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.7336, Chi-squared
Statistical Analysis 14: Comparison: Etanercept vs nbDMARDs; Leukaemia, Month 12: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.0044, Chi-squared
Statistical Analysis 15: Comparison: Etanercept vs nbDMARDs; Non-Melanoma Skin Cancer, Month 6: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.4175, Chi-squared
Statistical Analysis 16: Comparison: Etanercept vs nbDMARDs; Non-Melanoma Skin Cancer, Month 12: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.3886, Chi-squared
Statistical Analysis 17: Comparison: Etanercept vs nbDMARDs; Non-Melanoma Skin Cancer, Month 18: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.5102, Chi-squared
Statistical Analysis 18: Comparison: Etanercept vs nbDMARDs; Non-Melanoma Skin Cancer, Month 24: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.9855, Chi-squared
Statistical Analysis 19: Comparison: Etanercept vs nbDMARDs; Non-Melanoma Skin Cancer, Month 30: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.4955, Chi-squared
Statistical Analysis 20: Comparison: Etanercept vs nbDMARDs; Non-Melanoma Skin Cancer, Month 36: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.5404, Chi-squared
Statistical Analysis 21: Comparison: Etanercept vs nbDMARDs; Non-Melanoma Skin Cancer, Month 48: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.3581, Chi-squared
Statistical Analysis 22: Comparison: Etanercept vs nbDMARDs; Solid Tumor, Month 6: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.4932, Chi-squared
Statistical Analysis 23: Comparison: Etanercept vs nbDMARDs; Solid Tumor, Month 12: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.4818, Chi-squared
Statistical Analysis 24: Comparison: Etanercept vs nbDMARDs; Solid Tumor, Month 18: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.3224, Chi-squared
Statistical Analysis 25: Comparison: Etanercept vs nbDMARDs; Solid Tumor, Month 24: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.5003, Chi-squared
Statistical Analysis 26: Comparison: Etanercept vs nbDMARDs; Solid Tumor, Month 30: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.1134, Chi-squared
Statistical Analysis 27: Comparison: Etanercept vs nbDMARDs; Solid Tumor, Month 36: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.3488, Chi-squared
Statistical Analysis 28: Comparison: Etanercept vs nbDMARDs; Solid Tumor, Month 48: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.1870, Chi-squared
Statistical Analysis 29: Comparison: Etanercept vs nbDMARDs; Solid Tumor, Month 60: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.4270, Chi-squared

31. Other Pre Specified Outcome: Number of Participants Who Died or Hospitalized Due to Adverse Events
Description: Number of participants who died or hospitalized due to AEs is reported by each follow-up time point up to Month 60.
Time Frame: Month 6, 12, 18, 24, 30, 36, 48, 60
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 22 | 111
participants
  Death Due to AE: Month 6 (n=22, 101) | 1 | 8
  Death Due to AE: Month 12 (n=10, 100) | 1 | 3
  Death Due to AE: Month 18 (n=12, 111) | 0 | 3
  Death Due to AE: Month 24 (n=10, 102) | 2 | 2
  Death Due to AE: Month 30 (n=12, 80) | 0 | 0
  Death Due to AE: Month 36 (n=6, 91) | 0 | 2
  Death Due to AE: Month 48 (n=3, 63) | 0 | 0
  Death Due to AE: Month 60 (n=7, 44) | 1 | 6
  Hospitalization Due to AE: Month 6 (n= 18, 85) | 16 | 73
  Hospitalization Due to AE: Month 12 (n= 8, 81) | 6 | 70
  Hospitalization Due to AE: Month 18 (n= 11, 77) | 10 | 63
  Hospitalization Due to AE: Month 24 (n= 5, 70) | 5 | 62
  Hospitalization Due to AE: Month 30 (n= 8, 64) | 6 | 59
  Hospitalization Due to AE: Month 36 (n= 4, 69) | 4 | 59
  Hospitalization Due to AE: Month 48 (n= 1, 38) | 1 | 31
  Hospitalization Due to AE: Month 60 (n= 4, 24) | 4 | 22
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; Death Due to AE, Month 6: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.5817, Chi-squared
Statistical Analysis 2: Comparison: Etanercept vs nbDMARDs; Death Due to AE, Month 12: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.2595, Chi-squared
Statistical Analysis 3: Comparison: Etanercept vs nbDMARDs; Death Due to AE, Month 18: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.5642, Chi-squared
Statistical Analysis 4: Comparison: Etanercept vs nbDMARDs; Death Due to AE, Month 24: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.0034, Chi-squared
Statistical Analysis 5: Comparison: Etanercept vs nbDMARDs; Death Due to AE, Month 36: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.7137, Chi-squared
Statistical Analysis 6: Comparison: Etanercept vs nbDMARDs; Death Due to AE, Month 60: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.9630, Chi-squared
Statistical Analysis 7: Comparison: Etanercept vs nbDMARDs; Hospitalization Due to AE, Month 6: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.7353, Chi-squared
Statistical Analysis 8: Comparison: Etanercept vs nbDMARDs; Hospitalization Due to AE, Month 12: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.3829, Chi-squared
Statistical Analysis 9: Comparison: Etanercept vs nbDMARDs; Hospitalization Due to AE, Month 18: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.4532, Chi-squared
Statistical Analysis 10: Comparison: Etanercept vs nbDMARDs; Hospitalization Due to AE, Month 24: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.4238, Chi-squared
Statistical Analysis 11: Comparison: Etanercept vs nbDMARDs; Hospitalization Due to AE, Month 30: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.1218, Chi-squared
Statistical Analysis 12: Comparison: Etanercept vs nbDMARDs; Hospitalization Due to AE, Month 36: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.4124, Chi-squared
Statistical Analysis 13: Comparison: Etanercept vs nbDMARDs; Hospitalization Due to AE, Month 48: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.6356, Chi-squared
Statistical Analysis 14: Comparison: Etanercept vs nbDMARDs; Hospitalization Due to AE, Month 60: p-value was calculated using chi-square test; Test type: Superiority or Other; p = 0.5491, Chi-squared

32. Other Pre Specified Outcome: Change From Baseline in Disease Activity Score Based on 28-joints Count (DAS28) at Month 6
Description: DAS28 calculated from the SJC and PJC using the 28 joints count, acute phase reactants (ESR, millimeters per hour or CRP, milligram per liter) and PtGA of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). DAS28 <2.6: remission, DAS28 <=3.2: low disease activity, DAS28 >3.2 to <=5.1: moderate disease activity, DAS28 >5.1: progression.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 130 | 437
units on a scale | -0.63 (0.41) | 0.08 (0.39)
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; P-value was calculated using multivariate linear regression with baseline DAS28 score and other baseline variables (socio-demographics, disease characteristics, and initial treatment profile) as covariates; Test type: Superiority or Other; p < 0.0001, Regression, Linear

33. Other Pre Specified Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) Score at Month 6
Description: as for outcome 18
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 104 | 676
units on a scale | -0.14 (0.10) | 0.08 (0.09)
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; P-value was calculated using multivariate linear regression with baseline HAQ-DI score and other baseline variables (socio-demographics, disease characteristics, and initial treatment profile) as covariates; Test type: Superiority or Other; p < 0.0001, Regression, Linear

34. Other Pre Specified Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) at Month 6
Description: as for outcome 19
Time Frame: Baseline, Month 6
Population: as for outcome 9
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 104 | 711
units on a scale
  PCS (n= 87, 633) | 0.49 (1.40) | -0.34 (1.33)
  MCS (n= 87, 633) | -0.70 (1.42) | -1.21 (1.35)
  Vitality Score (n= 104, 711) | 1.84 (1.39) | 1.70 (1.33)
Statistical Analysis 1: Comparison: Etanercept vs nbDMARDs; PCS: p-value was calculated using multivariate linear regression with baseline PCS and other baseline variables (socio-demographics, disease characteristics, and initial treatment profile) as covariates; Test type: Superiority or Other; p = 0.2558, Regression, Linear
Statistical Analysis 2: Comparison: Etanercept vs nbDMARDs; MCS: p-value was calculated using multivariate linear regression with baseline MCS and other baseline variables (socio-demographics, disease characteristics, and initial treatment profile) as covariates; Test type: Superiority or Other; p = 0.4908, Regression, Linear
Statistical Analysis 3: Comparison: Etanercept vs nbDMARDs; Vitality Score: p-value was calculated using multivariate linear regression with baseline vitality score and other baseline variables (socio-demographics, disease characteristics, and initial treatment profile) as covariates; Test type: Superiority or Other; p = 0.8379, Regression, Linear

35. Other Pre Specified Outcome: Change From Baseline in Euro Quality of Life - 5 Dimensions (EQ-5D) at Month 6
Description: as for outcome 20
Time Frame: Baseline, Month 6
Population: Data not analyzed due to low number of participants available for this measure in BSRBR used for analysis.
Arm/Group | Etanercept | nbDMARDs
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: This study was a retrospective registry analysis of de-identified participants' data and only serious adverse events were available in the registry.
Arm/Group | Etanercept | nbDMARDs
Serious Adverse Events (participants affected / at risk) | 77/211 | 534/1543
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=211) | nbDMARDs (N=1543)
Pneumonia (General disorders) | 3 | 63
Septicaemia (General disorders) | 0 | 5
Bone/Joint Infection (General disorders) | 2 | 5
Other Infection (General disorders) | 13 | 40
Congestive Heart Failure (General disorders) | 1 | 7
Myocardial Infarction (General disorders) | 3 | 19
Other Cardiac Events (General disorders) | 2 | 31
Central Demyelination (General disorders) | 0 | 1
Optic Neuritis (General disorders) | 1 | 0
Peripheral Neuropathy (General disorders) | 0 | 5
Other CNS Events (General disorders) | 8 | 30
Pancytopaenia (General disorders) | 0 | 2
Leukopaenia (General disorders) | 0 | 2
Other Dyscrasia (General disorders) | 0 | 16
Lymphoproliferative Tumors (General disorders) | 5 | 6
Hodgkin's Lymphoma (General disorders) | 4 | 4
Myeloma (General disorders) | 0 | 2
Leukaemia (General disorders) | 1 | 0
Non-Melanoma Skin Cancer (General disorders) | 1 | 30
Solid Tumor (General disorders) | 6 | 46
Other Infection (General disorders) | 16 | 109
Tuberculosis (TB) (General disorders) | 0 | 1
Pregnancy (General disorders) | 5 | 6
Other Serious Events (General disorders) | 30 | 422

LIMITATIONS AND CAVEATS:
Since this study was a retrospective registry analysis of de-identified participants' data, only SAEs pre specified in analysis were reported with preferred terms and all other SAEs were reported under the preferred term Other Serious Event.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.